CLINICAL TRIAL: NCT00372203
Title: Prospective Controlled Trial of Mediastinoscopy Compared With Endobronchial Ultrasound Guided Transbronchial Needle Aspiration for Assessment of the Mediastinum in Lung Cancer.
Brief Title: Endobronchial Ultrasound vs Mediastinoscopy in NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 06-0085-A
Record Dates: First submitted 2006-09-04; First posted 2006-09-06 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; NSCLC; EBUS; Endobronchial ultrasound; mediastinoscopy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endobronchial ultrasound (Experimental)
  Interventions: Procedure: Endobronchial Ultrasound Guided Transthoracic Needle Biopsy

INTERVENTIONS:
Procedure: Endobronchial Ultrasound Guided Transthoracic Needle Biopsy — Endobronchial Ultrasound Guided Transthoracic Needle Biopsy of mediastinal lymph nodes at the time of the mediastinoscopy.

SUMMARY:
Proper staging of Lung cancer is of paramount concern when determining a treatment regime. Currently the assessment of surgical candidacy is performed with the staging process, mainly the mediastinoscopy. A mediastinoscopy has the ability to access samples of the paratracheal lymph node stations (Levels 2R, 2L, 3, 4R, 4L), as well as the anterior subcarinal lymph node station (Level 7). In comparison, the EBUS-TBNA technique is a real-time procedure that has the potential to access the same paratracheal and subcarinal lymph node stations associated with the mediastinoscopy, but also extending out to the hilar lymph nodes (Levels 10 and 11). Because of the possibility of extended sampling range and a reduction in procedural invasiveness, EBUS-TBNA may represent a more efficient patient centered alternative to mediastinoscopy in the staging of lung cancer patients. Additionally, patients who are have lymph nodes in the N2 region frequently undergo chemotherapy and/or radiotherapy prior to surgery. Assessment of the lymph nodes after chemo/radiation is done using CT scans, as re-mediastinoscopy is a technically difficult procedure. These patients may benefit from EBUS-TBNA.

ELIGIBILITY:
Inclusion Criteria:

A) Age 18 years or older B) Patients with confirmed or suspected non-small cell lung cancer who require a mediastinoscopy as part of their staging investigations of the mediastinum to determine suitability for lung cancer resection will be considered for the trial.

C) Patients with undiagnosed enlarged lymph nodes in the mediastinum suspicious for lung cancer in which a tissue diagnosis is required.

Exclusion Criteria:

A) Patients who are deemed on clinical grounds not to be medically fit for a bronchoscopy or a mediastinoscopy or who are not suitable for definitive surgical resection by thoracotomy will be excluded.

B) Patients who have verified stage IV disease or who are not appropriate for lung cancer resection by virtue of direct invasion of mediastinal structures or large parts of the chest wall.

C) Known small cell lung cancer. D) Patients where there is a high clinical suspicion of lymphoma. E) Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Sensitivity | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Shaf Keshavjee, MD MSc FRCSC FACS, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network (Toronto General Hospital), Toronto, Ontario, Canada